CLINICAL TRIAL: NCT00948480
Title: Vaccine Biotherapy Of Cancer: Autologous Tumor Cells and Dendritic Cells as Active Specific Immunotherapy in Patients With Metastatic Melanoma
Brief Title: Vaccine Biotherapy of Cancer: Autologous Tumor Cells and Dendritic Cells
Acronym: DCVaccineMel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC Melanoma
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Metastatic Melanoma
Keywords: autologous tumor cell vaccine; metastatic melanoma; sargramostim (GM-CSF)
MeSH Terms: conditions — Melanoma | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Autologous tumor cells plus dendritic cells — A series of 8 vaccinations are administered over 6 months
Drug: GM-CSF — 500 mcg
  Other Names: Sargramostim

SUMMARY:
This protocol was conducted as a single institution trial at Hoag Cancer Center, Hoag Hospital, Newport Beach, California. It was a single-arm phase II trial in which patients with metastatic melanoma received subcutaneous (s.c.) injections of irradiated autologous tumor cells that had been established as short-term cell lines, in conjunction with their own dendritic cells (DC) and granulocyte macrophage colony-stimulating factor [GM-CSF]. Eligible patients had regionally recurrent and/or distant metastatic cancer.

DETAILED DESCRIPTION:
Patients were stratified by whether they had no measurable disease [NMD] at the time of treatment (usually because of surgical resection of metastases), or whether they had objectively measurable disease (OMD) by physical examination or radiologic scans per response evaluation criteria in solid tumors (RECIST criteria). Key endpoints were the results of delayed type hypersensitivity (DTH) skin testing to their own irradiated tumor cells, event-free survival [death or disease progression], overall survival, and objective tumor regression in patients who have measurable disease at the time vaccine therapy was initiated. This study was activated in the fall of 2000, and closed to accrual in June 2007.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or metastatic melanoma as defined by stage IV disease (distant metastases), or any recurrent melanoma manifested by lymph node metastases or soft tissue nodules
* ECOG Performance status of 0-2
* Satisfactory medical condition for treatment in a phase I-II trial of anticancer therapy
* Age > 16 years
* Venous access for leukopheresis procedure to obtain peripheral blood lymphocytes to generate dendritic cells.
* Serum pregnancy test must be negative for women of childbearing potential.

Exclusion Criteria:

* Active central nervous system metastases
* Known autoimmune disease or disease process that involves the use of immunosuppressive therapy.
* Underlying cardiac disease associated with New York Heart Association class III or IV function, or unstable angina related to atherosclerotic cardiovascular disease.
* Ongoing transfusion requirements, no significant hepatic or renal dysfunction, creatinine < 2.0 mg/dl, bilirubin < 2.0 mg/dl, albumin > 3.0 mg/dl, hematocrit > 25, platelets > 100,000.
* Active infection or other active medical condition that could be eminently life threatening, including no active blood clotting or bleeding diathesis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2000-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
event-free survival [death or disease progression] | 5.5 years after treatment initation

SECONDARY OUTCOMES:
Overall survival | 5.5 years after treatment initation

CONTACTS AND LOCATIONS:
Overall Officials: Robert O Dillman, MD, Principal Investigator — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

REFERENCES:
- [Result] Dillman RO, Selvan SR, Schiltz PM, McClay EF, Barth NM, DePriest C, de Leon C, Mayorga C, Cornforth AN, Allen K. Phase II trial of dendritic cells loaded with antigens from self-renewing, proliferating autologous tumor cells as patient-specific antitumor vaccines in patients with metastatic melanoma: final report. Cancer Biother Radiopharm. 2009 Jun;24(3):311-9. doi: 10.1089/cbr.2008.0599. PMID 19538053
- [Derived] Dillman RO, Cornforth AN, McClay EF, Depriest C. Patient-specific dendritic cell vaccines with autologous tumor antigens in 72 patients with metastatic melanoma. Melanoma Manag. 2019 May 31;6(2):MMT20. doi: 10.2217/mmt-2018-0010. PMID 31406564
- [Derived] Dillman RO, Cornforth AN, Nistor GI, McClay EF, Amatruda TT, Depriest C. Randomized phase II trial of autologous dendritic cell vaccines versus autologous tumor cell vaccines in metastatic melanoma: 5-year follow up and additional analyses. J Immunother Cancer. 2018 Mar 6;6(1):19. doi: 10.1186/s40425-018-0330-1. PMID 29510745